CLINICAL TRIAL: NCT01370135
Title: An Open Label, Prospective, Monocenter, Prove of Concept Study to Evaluate the Short- and Long-term Effects of 0.5mg Intraocular Ranibizumab (Lucentis) Injections as Adjuvant for Patients With Rubeosis and Neovascular Glaucoma
Brief Title: Study to Evaluate the Effects of Ranibizumab (Lucentis) for Patients With Rubeosis and Neovascular Glaucoma
Acronym: LucNVG0108
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Luebeck (Other)
Responsible Party: Principal Investigator, Dr. Julia Lueke, Dr. med. Julia Lüke, University of Luebeck
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LucNVG0108
Record Dates: First submitted 2011-05-27; First posted 2011-06-09 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Neovascular Glaucoma; Rubeosis
Keywords: neovascular glaucoma; rubeosis; anterior chamber; intraocular; intravitreal injections; Lucentis; Ranibizumab; short ans longterm effects; best corrected visual acuity; gonioscopy; BCVA; quality of life
MeSH Terms: conditions — Glaucoma, Neovascular | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lucentis (Ranibizumab) (Experimental)
  Interventions: Drug: 0.5mg intraocular Ranibizumab (Lucentis)

INTERVENTIONS:
Drug: 0.5mg intraocular Ranibizumab (Lucentis) — short- and long-term effects of 0.5mg intraocular Ranibizumab (Lucentis) injections as adjuvant for patients with rubeosis and neovascular glaucoma

SUMMARY:
Proliferative ischemic retinopathies lead to a formation of abnormal vessels on the iris surface induced by an increased level of vascular endothelial growth factor (VEGF). In progressive stages fibrovascular membranes occlude the anterior chamber angle which inhibits aqueous outflow resulting in neovascular glaucoma. The increased intraocular pressure is often difficult to control and frequently results in loss of vision.

The aim of this study is to analyze the short- and long-term outcome after adjuvant intraocular Ranibizumab application in patients with neovascular glaucoma and rubeosis and to analyze the role of ranibizumab within a holistic treatment regime.

ELIGIBILITY:
Inclusion Criteria:

1. neo-vascular glaucoma or rubeosis

   * definition of neo-vascular glaucoma: patient with iris neovascularization with intraocular pressure elevation (exceeding 21 mmHg)
   * definition of rubeosis: patient with iris neovascularization without intraocular pressure elevation (≤21 mmHg)
2. an available follow-up of 12 months
3. written informed consent
4. visual acuity of light perception or better.

Exclusion Criteria:

1. history or evidence of severe cardiac disease (e.g., NYHA functional class III or IV)
2. clinical or medical history of unstable angina, acute coronary syndrome, myocardial infarction or revascularization with 6 months
3. ventricular tachyarrhythmias requiring ongoing treatment
4. History or evidence clinically significant peripheral vascular disease, such as intermittent claudication or prior amputation
5. Clinically significant impaired renal or hepatic function
6. Stroke within 12 month before trial entry.
7. Known serious allergies to the fluorescein dye use in angiography
8. Known contraindications to the components of Lucentis® formulation.

Ocular concomitant conditions/ diseases

1. Active intraocular inflammation (grade trace or above) in either eye
2. Any active infection (e.g. conjunctivitis, keratitis, scleritis, uveitis, endophthalmitis) in either eye
3. History of uveitis in either eye
4. Treatment with anti-angiogenic drugs (pegaptanib sodium, anecortave acetate,bevacizumab, ranibizumab, etc.) or intravitreal corticosteroids in either eye within 4 months prior to inclusion
5. Angle block glaucoma
6. Phthisis
7. Intraocular Pressure <10mmHg

Compliance/ Administrative

1. Previous participation in any clinical studies of investigational drugs (excluding vitamins and minerals) within 1 month (or a period corresponding to 5 half-lives of the investigational drug, whatever is longer) prior to inclusion
2. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant. including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS they are using two birth control methods. The two methods can be a double barrier method or a barrier method plus a hormonal method. Adequate barrier methods of contraception include: diaphragm, condom (by the partner), intrauterine device (copper or hormonal), sponge or spermicide. Hormonal contraceptives include any marketed contraceptive agent that includes an estrogen and/or a progestational agent.
3. Pregnant or nursing (lactating) women
4. Inability to comply with study or follow-up procedures.
5. Any treatment with an investigational agent in the past 60 days for any condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-11; Primary Completion 2011-04 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
change of degree of iris rubeosis | 12 Months
  Main outcome measure is the change of degree of iris rubeosis as documented by iris fluorescein angiography as measured 12 months after the first ranibizumab injection.

SECONDARY OUTCOMES:
changes in intraocular pressure | 12 Months
  • to document changes in intraocular pressure measurements with the Goldmann applanation tonometer
changes in best corrected visual acuity (BCVA) | 12 Months
  • to document changes in best corrected visual acuity (BCVA) measured on 4 meters
numbers of additional interventions | 12 Months
  • to document numbers of additional interventions or anti-glaucomatous medications 12 months after injection
quality of life | 12 Months
  • to document changes of quality of life
Number of adverse events in all participants | 12 Months
  • to evaluate the safety of intravitreal injections of ranibizumab (0.5 mg) as adjunctive in patients with rubeosis and neovascular glaucoma using the number of adverse events.
changes in gonioscopy | 12 Months
  • to document changes in gonioscopy of the anterior chamber angle

CONTACTS AND LOCATIONS:
Overall Officials: Salvatore Grisanti, M.D. Prof., Principal Investigator — University of Lübeck - Department of Ophthalmology: Germany
Locations (1):
- University of Lübeck - Department of Ophthalmology, Lübeck, Germany

REFERENCES:
- [Derived] Luke J, Nassar K, Luke M, Grisanti S. Ranibizumab as adjuvant in the treatment of rubeosis iridis and neovascular glaucoma--results from a prospective interventional case series. Graefes Arch Clin Exp Ophthalmol. 2013 Oct;251(10):2403-13. doi: 10.1007/s00417-013-2428-y. Epub 2013 Jul 28. PMID 23893090
- See also: University of Lübeck - Department of Ophthalmology - Germany — http://www.uksh.de/Augenklinik_Luebeck/index.html